CLINICAL TRIAL: NCT06701565
Title: Coronal and Radicular Caries Prevalence With Related Risk Factors Among Middle Age Type II Diabetic Patients Attending National Institute of Diabetes and Endocrinology: a Hospital Based Cross Sectional Study
Brief Title: Coronal and Radicular Caries Prevalence and Related Risk Factor in Diabetic Patient
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Osama Rashid, principal investigator, Cairo University
Other Study IDs: Caries Prevalence and Diabetes
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Caries,Dental; Caries Root; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Dental Caries; Root Caries; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controlled type 2 diabetes
- Uncontrolled type 2 diabetes

SUMMARY:
This study aims to investigate the prevalence and risk factors of coronal and radicular caries in middle-aged individuals with Type 2 diabetes. It focuses on how poor blood sugar control, reduced saliva production, increased plaque accumulation, and periodontal disease contribute to a higher risk of dental decay in this population. The study examines the relationship between glycemic control (e.g., HbA1c levels) and the severity of caries, as well as the impact of diabetes-related changes in oral health, such as gum recession and dry mouth, on the development of both coronal and radicular caries. The findings could inform preventive strategies and dental care guidelines tailored for diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient whose age between 30-65
2. Diabetic patients
3. Patient consulting in the outpatient clinic
4. Co-operative patient
5. Males & Females
6. Egyptian

Exclusion Criteria:

1. Patients under or over this age group
2. Lack of compliance
3. Disabilities
4. Pregnant women

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1. Patient whose age between 30-65
  2. Diabetic patients
  3. Patient consulting in the outpatient clinic
  4. Co-operative patient
  5. Males & Females
  6. Egyptian
Sampling Method: Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
prevalence of coronal caries | One year
  DMFT Index developed by World Health Organization (WHO) using number scores and percentage
prevalence of radicular caries | One year
  Radicular caries by International Caries and Assessment System (ICDAS II)

SECONDARY OUTCOMES:
Blood Glucose level | One year
  Blood tests of glycated hemoglobin
Salivary flow | One year
  Graduated test tube
Salivary pH | One year
  PH indicator
Caries risk related factors | one year
  WHO oral health questionnaire for adults 2013